CLINICAL TRIAL: NCT01085942
Title: Longitudinal Study of Asymptomatic Rotator Cuff Tears. A Eight Year Follow-up of Symptomatic Status and Tear Characteristics Like Tear Size, Muscle Atrophy and Fatty Degeneration
Brief Title: Longitudinal Study of Asymptomatic Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Stefan Moosmayer, MD, PhD, Vestre Viken Hospital Trust
Other Study IDs: 288-05082 (REK); 2006049 (Other: Helse Soer-Oest)
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff tear; asymptomatic; natural course; tear characteristics; Asymptomatic rotator cuff tears; Natural course of rotator cuff tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asymptomatic rotator cuff tear: Subjects identified with an asymptomatic rotator cuff tear

SUMMARY:
The purpose of this study is to analyze the natural course of asymptomatic rotator cuff tears.

DETAILED DESCRIPTION:
Fifty subjects with an asymptomatic rotator cuff tear were identified in an earlier study. Clinical, sonographic and MRI reexamination of these subjects is performed after an interval of three years. Findings of interest include: (1) the symptomatic status of the subjects (still asymptomatic or symptomatic); (2)tear size on sonography and MRI (unchanged or increased); (3)degree of muscle atrophy on MRI (unchanged or deteriorated); (4)degree of fatty muscle degeneration on MRI (unchanged or deteriorated). We want to analyze whether a change in these tear characteristics is associated with a change of the symptomatic status of these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an asymptomatic rotator cuff tear at least in one shoulder, tear demonstrated both on MRI and sonography, ASES score exceeding 90 points

Exclusion Criteria:

* Earlier periods with shoulder pain and dysfunction, earlier treatment for shoulder problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects identified with an asymptomatic rotator cuff tear
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Symptoms from a rotator cuff tear | 8 years
  The symptomatic status of initially asymptomatic rotator cuff tears is followed up by reexamination after three and eight years
Tear characteristics on MRI and sonography | 8 years
  Tear characteristics from initially asymptomatic rotator cuff tears are followed up by reexamination by MRI and sonography after three and eight years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Moosmayer, MD, Principal Investigator — Vestre Viken Hospital Trust
Locations (1):
- Martina Hansen's Hospital, Sandvika, Norway

REFERENCES:
- [Background] Keener JD. Surveillance of conservatively treated rotator cuff tears is warranted. Commentary on an article by Stefan Moosmayer, MD, PhD, et al.: "The natural history of asymptomatic rotator cuff tears. a three-year follow-up of fifty cases". J Bone Joint Surg Am. 2013 Jul 17;95(14):e101 1-2. doi: 10.2106/JBJS.M.00526. No abstract available. PMID 23864184
- [Result] Moosmayer S, Smith HJ, Tariq R, Larmo A. Prevalence and characteristics of asymptomatic tears of the rotator cuff: an ultrasonographic and clinical study. J Bone Joint Surg Br. 2009 Feb;91(2):196-200. doi: 10.1302/0301-620X.91B2.21069. PMID 19190053
- [Result] Moosmayer S, Tariq R, Stiris MG, Smith HJ. MRI of symptomatic and asymptomatic full-thickness rotator cuff tears. A comparison of findings in 100 subjects. Acta Orthop. 2010 Jun;81(3):361-6. doi: 10.3109/17453674.2010.483993. PMID 20450423
- [Result] Moosmayer S, Tariq R, Stiris M, Smith HJ. The natural history of asymptomatic rotator cuff tears: a three-year follow-up of fifty cases. J Bone Joint Surg Am. 2013 Jul 17;95(14):1249-55. doi: 10.2106/JBJS.L.00185. PMID 23864172